CLINICAL TRIAL: NCT03818737
Title: Randomized Multicenter Phase 3 Single-blind Trial Comparing the Efficacy of Corticosteroid Control to Mesenchymal Stem Cell Preparations From Autologous Bone Marrow Concentrate (BMAC), Adipose-derived Stem Cells in the Form of Stromal Vascular Fraction (SVF), and Third-party Human Mesenchymal Stem Cells Manufactured From Umbilical Cord Tissue for the Treatment of Unilateral Knee Osteoarthritis (OA)
Brief Title: Multicenter Trial of Stem Cell Therapy for Osteoarthritis (MILES)
Acronym: MILES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, Scott D Boden, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00108046
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis
Keywords: mesenchymal stem cells; corticosteroids; bone marrow aspiration; adipose-derived stromal vascular fraction
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones; Methylprednisolone Acetate; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: The study will include a parallel design using a blocked central randomization scheme of 1:1:1:1. Participants will first be randomized to have MSCs derived from either bone marrow, adipose tissue, or umbilical cord tissue. Then they will be further randomized to receive either an injection of MSCs (from bone marrow, adipose, or umbilical cord tissue, depending on the first randomization) or a corticosteroid injection.
Who Masked: Participant
Masking Description: Participants will not know if they are receiving the MSC or corticosteroid injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Bone Marrow Derived MSCs (Experimental): Participants randomized to this arm will undergo bone marrow aspiration and then will be further randomized to receive a standard orthobiologic injection into the knee joint of autologous bone marrow concentrate (BMAC).
  Interventions: Biological: Bone Marrow Derived MSCs
- Adipose-derived MSCs (Experimental): Participants randomized to this arm will undergo small volume lipoplasty, and then will be further randomized to receive an injection into the knee joint of adipose-derived stromal vascular fraction (SVF).
  Interventions: Biological: Adipose-derived MSCs
- Umbilical Cord Tissue (UCT) MSCs (Experimental): Participants randomized to this arm will receive an injection into the knee joint of cryopreserved doses of umbilical cord tissue MSCs.
  Interventions: Biological: Umbilical Cord Tissue (UCT) MSCs
- Corticosteroid Injection (Active Comparator): Participants randomized to the bone marrow derived MSC, adipose-derived MSC, or umbilical cord tissue MSC study arms will be further randomized within the arm in a 3:1 ratio to receive either MSCs derived from the study arm of the initial randomization or a corticosteroid (CS) injection. Participants randomized to the control group will receive an injection of corticosteroid into the knee joint.
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Biological: Bone Marrow Derived MSCs — Autologous bone marrow concentrate (BMAC) is a standard orthobiologic injection for knee osteoarthritis. The procedure involves harvesting of bone marrow aspirate (BMA) from the posterior superior iliac spine (PSIS) and then following centrifugation in an FDA approved device (EmCyte GenesisCS Pure BMAC®-60 ml) will be injected back into the knee joint. All injections will be made via ultrasound guidance using a standard approach.
  Arms: Bone Marrow Derived MSCs
Biological: Adipose-derived MSCs — Adipose-derived Stromal Vascular Fraction (SVF) will be obtained from a mini lipoaspirate. The lipoaspirate will then be enzymatically digested to produce a SVF that will be injected into the knee joint. All injections will be made via ultrasound guidance using a standard approach.
  Arms: Adipose-derived MSCs
Biological: Umbilical Cord Tissue (UCT) MSCs — Cryopreserved doses of umbilical cord tissue MSCs will be used. These MSCs were cryopreserved at P2 culture in plasmalyte A + 5% human serum albumin in 5 finger cryobags containing 20 million cells in 4 mL and stored under liquid nitrogen until shipment. Cells will be transported in a dry shipper and thawed at the study sites. The dose of MSCs will be aspirated from the cryobag into a sterile syringe and directly injected into the knee. All injections will be made via ultrasound guidance using a standard approach.
  Arms: Umbilical Cord Tissue (UCT) MSCs
Drug: Corticosteroid injection — The corticosteroid injection is prepared by mixing 1cc of 40mg/dL depomedrol and 6cc of normal saline in a 10cc syringe will be made into the knee joint. All injections will be made via ultrasound guidance using a standard approach.
  Other Names: Depo-Medrol; Methylprednisolone
  Arms: Corticosteroid Injection

SUMMARY:
The study is a multicenter trial conducted to compare the effectiveness of an injection of a corticosteroid control to mesenchymal stem cell (MSC) preparations from autologous bone marrow concentrate (BMAC), adipose derived stem cells in the form of Stromal Vascular Fraction (SVF), and third-party human mesenchymal stem cells manufactured from umbilical cord tissue (UCT) for the treatment of unilateral Knee Osteoarthritis (OA). The study will be conducted in 4 sites in the United States, and a total of 480 participants will be enrolled in this study.

DETAILED DESCRIPTION:
Primary osteoarthritis is a debilitating disease characterized by extensive damage to the joints and excruciating pain leading to loss of activity and depression. Despite advances in diagnosis and relatively efficient control of nociception, to date, the quest for the development of a disease modifying osteoarthritis drug has proven unsuccessful. The potential of mesenchymal stem cells (MSCs) to inhibit inflammation while promoting healing makes them amenable for the treatment of various ailments ranging from cancer to genetic diseases. In orthopedic practice, autologous stem cell injections are performed to alleviate the pain associated with osteoarthritis. A serious gap in knowledge remains whether the currently used cellular treatments are beneficial in the long term and if one cell therapy outperforms another.

The most popular form of autologous MSC therapy has been through the use of autologous bone marrow concentrate (BMAC). The rationale is that when a sample of bone marrow aspirate (BMA) is collected and the components that are not beneficial to the joint are filtered out (i.e. red blood cells, neutrophils, etc.) the remaining concentrate (MSCs, platelets, interleukins, etc) can have a "healing" effect on the environment in which it is injected. However it is still unknown as to how effective BMAC is for treating orthopedic conditions compared to other MSC procedures and the most important components of the BMAC mixture that could aid patients suffering from osteoarthritis.

Adipose tissue has been found to have a large amount of MSCs versus that in bone marrow. These cells are currently being used in a variety of clinical research studies within the regenerative medicine field. Through a tissue process which includes washing and centrifuging, the cellular components can be extracted as a cell pellet, which is also known as stromal vascular fraction (SVF). Adipose derived SVF is obtained via liposuction, or the removal of adipose tissue via a suction method.

Although the use of various stem cell preparations for knee osteoarthritis has become increasingly prevalent, well-designed studies with conclusive proof of comparative effectiveness and identification of the optimal cell source and "dose" have not been performed. This study is the first randomized study comparing three types of cellular treatments to corticosteroids. The main objective of the study is to identify a superior source of stem cells for the treatment of osteoarthritis and validate its advantages over corticosteroid injections as the traditional gold standard treatment.

Participants will be randomized study arms with different types of MSCs (bone marrow derived MSC, adipose derived MSC, and umbilical cord tissue MSC) and then will be further randomized to receive an injection of the MSC type they were initially assigned to or corticosteroid. Participants randomized to bone marrow derived MSC or adipose derived MSC will undergo a procedure (bone marrow aspiration or liposuction). Participants will be blinded to whether they receive the MSC or corticosteroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 40 but less than or equal to 70 years old
* Males and females
* Recent knee radiograph of the targeted knee (standing anteroposterior (AP) lateral and sunrise view)
* Diagnosis of OA in the targeted knee (radiographic evidence of OA in the medial and/or lateral tibiofemoral compartment, which would include one or more osteophytes on a standard radiograph taken within 3 months)
* Continued OA pain in the targeted knee despite conservative measures (per treating provider's discretion)
* Average daily Visual Analog Scale (VAS) ≥3
* Kellgren-Lawrence system of Grade II, III, or IV
* Subjects may have concomitant patellofemoral but they must have stage II or higher generalized knee OA
* Females of childbearing potential only, must have a negative pregnancy test done at screening prior to enrollment in the study
* Women and men of child-producing potential must agree to use acceptable contraception methods for the duration of the trial such as birth control pills or condoms with spermicide

Exclusion Criteria:

* Clinically apparent tense effusion of the targeted knee
* Significant valgus/varus deformities (+/- 10 degrees)
* Viscosupplementation within 6 months in the targeted knee
* Other biologic injection (PRP or stem cell) within 1 year in the targeted knee
* Surgery in the targeted knee within the past 6 months (either open or scope)
* Systemic or intra-articular injection of corticosteroids in any joint within 3 months before screening
* Daily opioid use for the past three months
* History of malignancy in the previous 5 years prior to study entry, with the exception of in-situ cancers treated only by local excision with curative intent
* History of, or ongoing, autoimmune disorder that requires treatment with an immunosuppressive medication
* Active, suspected, or prior infection to the joint in the targeted knee
* Part of a vulnerable population per Office for Human Research Protections (OHRP) definition (pregnant women and breast-feeding women, cognitively impaired, prisoners, etc.)
* Unwilling to discontinue the use of Non-Steroidal Anti-Inflammatory (NSAID)s for 7 calendar days prior to the procedure
* Unwilling to discontinue use of NSAIDS for 5 calendar days after procedure
* History of bleeding disorders or inflammatory joint disease
* Inability to hold anti-platelet therapy according to treating provider prior to procedure
* Subject is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason
* Uncontrolled diabetes
* Subject has an active workers' compensation case in progress with targeted knee
* Subject with insufficient amount of subcutaneous tissue
* Hemoglobin less than 10g/dL at the time of screening
* Leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL at the time of screening
* Diagnosis of liver disease as defined by alanine aminotransferase (ALT) >3x the upper limit of age-determined normal (ULN) or total bilirubin > 1.5x ULN
* Subjects who have had greater than 3 corticosteroid injections in the targeted knee in the 12 months prior to screening or at the physician's discretion
* Subjects with a known diagnosis of osteoporosis
* Subjects with anticipated use of systemic corticosteroids during the study period for treatment of a chronic medical condition

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hicham Drissi, PhD, Study Director — Emory University; Scott D Boden, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Andrews Institute, Gulf Breeze, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Duke University, Durham, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mautner K, Kaiser JM, Boggess B, Hackel J, Kurtenbach C, Noonan B, Shenvi N, Easley KA, Myer GD, Jayaram P, Gottschalk M, Boden S, Drissi H. Autologous Cell Injections for Knee Osteoarthritis Display Greater Responsiveness Than Allogenic Cellular Products and Corticosteroids in a Sex-Dependent Manner. Am J Sports Med. 2025 Oct;53(12):2889-2897. doi: 10.1177/03635465251365521. Epub 2025 Sep 27. PMID 41014273
- [Derived] Mautner K, Gottschalk M, Boden SD, Akard A, Bae WC, Black L, Boggess B, Chatterjee P, Chung CB, Easley KA, Gibson G, Hackel J, Jensen K, Kippner L, Kurtenbach C, Kurtzberg J, Mason RA, Noonan B, Roy K, Valentine V, Yeago C, Drissi H. Cell-based versus corticosteroid injections for knee pain in osteoarthritis: a randomized phase 3 trial. Nat Med. 2023 Dec;29(12):3120-3126. doi: 10.1038/s41591-023-02632-w. Epub 2023 Nov 2. PMID 37919438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Duke University in Durham, North Carolina, Sanford Health in Fargo, North Dakota, The Emory Clinic in Atlanta, Georgia, Sanford Health in Sioux Falls, South Dakota, and the Andrews Institute in Gulf Breeze, Florida, USA. Participant enrollment began March 28, 2019 and all follow-up was complete by May 31, 2022.
Groups:
- Bone Marrow Derived Mesenchymal Stem Cells (MSCs): Participants randomized to this arm underwent bone marrow aspiration and then were further randomized to receive a standard orthobiologic injection into the knee joint of autologous bone marrow concentrate (BMAC).
- Adipose-derived MSCs: Participants randomized to this arm underwent small volume lipoplasty, and then were further randomized to receive an injection into the knee joint of adipose-derived stromal vascular fraction (SVF).
- Umbilical Cord Tissue (UCT) MSCs: Participants randomized to this arm received an injection into the knee joint of cryopreserved doses of umbilical cord tissue MSCs.
- Corticosteroid Injection: Participants randomized to the bone marrow derived MSCs, adipose-derived MSCs, or umbilical cord tissue MSCs study arms who were further randomized to the control group and received a corticosteroid (CS) injection into the knee joint.
Period: Overall Study
Arm/Group | Bone Marrow Derived Mesenchymal Stem Cells (MSCs) | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Started (Intent to treat population) | 118 | 119 | 118 | 120
Received Study Intervention | 107 | 109 | 116 | 108
Completed | 97 | 93 | 103 | 97
Not Completed | 21 | 26 | 15 | 23

BASELINE CHARACTERISTICS:
Groups:
- Bone Marrow Derived MSCs: Participants randomized to this arm underwent bone marrow aspiration and then were further randomized to receive a standard orthobiologic injection into the knee joint of autologous bone marrow concentrate (BMAC).
- Corticosteroid Injection: Participants randomized to the bone marrow derived MSC, adipose-derived MSC, or umbilical cord tissue MSC study arms who were further randomized to the control group and received a corticosteroid (CS) injection into the knee joint.
- Total: Total of all reporting groups
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection | Total
Number analyzed (Participants) | 118 | 119 | 118 | 120 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.33) | 58.2 (7.31) | 57.9 (8.18) | 58.3 (8.05) | 58.3 (7.71)
Age, Customized [Count of Participants; unit: Participants]
  Categorical age: 40 to 59 years of age | 57 | 63 | 64 | 62 | 246
  Categorical age: 60 to 70 years of age | 61 | 56 | 54 | 58 | 229
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 63 | 65 | 71 | 261
  Male | 56 | 56 | 53 | 49 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5 | 6 | 16
  Not Hispanic or Latino | 116 | 113 | 113 | 114 | 456
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 4 | 3 | 4 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 15 | 11 | 12 | 57
  White | 92 | 99 | 102 | 104 | 397
  More than one race | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118 | 119 | 118 | 120 | 475

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Pain Scale (VAS-pain) Score
Description: Pain assessment was performed using the Visual Analog Pain Scale (VAS-pain). The VAS-pain is self-completed by the participant. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance in millimeters (mm) on the line between the "no pain" anchor and the participant's mark, providing a range of scores from 0-100. The recommended cut points for VAS are: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). The change in VAS-pain score is the score from the each follow-up visit subtracted from the baseline score. A negative value means that pain has reduced from what it was at baseline.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: This analysis includes participants who successfully completed this assessment at the indicated post-baseline study visit. Some participants withdrew from the study prior to study completion and some attended study visits but did not complete each study assessment correctly.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 101 | 102 | 111 | 101
units on a scale
  Absolute Change from Baseline at Month 1: number analyzed (Participants) | 101 | 101 | 111 | 101
  Absolute Change from Baseline at Month 1 | -20.2 (2.52) | -15.9 (2.48) | -16.7 (2.40) | -25.2 (2.49)
  Absolute Change from Baseline at Month 3: number analyzed (Participants) | 98 | 102 | 105 | 101
  Absolute Change from Baseline at Month 3 | -28.8 (2.54) | -17.8 (2.48) | -17.3 (2.43) | -21.1 (2.49)
  Absolute Change from Baseline at Month 6: number analyzed (Participants) | 94 | 94 | 99 | 97
  Absolute Change from Baseline at Month 6 | -23.2 (2.56) | -21.6 (2.53) | -19.7 (2.47) | -22.7 (2.51)
  Absolute Change from Baseline at Month 9: number analyzed (Participants) | 83 | 81 | 83 | 81
  Absolute Change from Baseline at Month 9 | -21.9 (2.64) | -17.9 (2.63) | -16.5 (2.58) | -23.3 (2.63)
  Absolute Change from Baseline at Month 12: number analyzed (Participants) | 95 | 91 | 98 | 97
  Absolute Change from Baseline at Month 12 | -25.5 (2.56) | -19.9 (2.55) | -20.6 (2.48) | -22.3 (2.51)

2. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) - Pain Subscale Score
Description: The KOOS questionnaire assesses the participant's opinion about their osteoarthritis and associated problems. It consists of 5 subscales: pain, symptoms, activities of daily living (ADL) function, sport and recreation function, and knee related quality of life (QoL). The pain subscale has 9 items and response options are given on a 5-point Likert scale where 0 = no problems and 4 = extreme problems. Scores are transformed to a scale ranging from 0 to 100 with 0 indicating extreme symptoms and 100 indicating no symptoms. The change in KOOS-pain subscale score is the score from each follow-up visit subtracted from the baseline score. A negative value means that pain has worsened from what it was at baseline, while a positive value means that pain has improved from baseline.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 101 | 101 | 111 | 101
score on a scale
  Absolute Change from Baseline at Month 1: number analyzed (Participants) | 101 | 100 | 111 | 101
  Absolute Change from Baseline at Month 1 | 15.5 (1.85) | 15.4 (1.84) | 11.5 (1.77) | 19.2 (1.83)
  Absolute Change from Baseline at Month 3: number analyzed (Participants) | 99 | 101 | 105 | 101
  Absolute Change from Baseline at Month 3 | 19.2 (1.86) | 16.8 (1.84) | 12.8 (1.79) | 18.7 (1.83)
  Absolute Change from Baseline at Month 6: number analyzed (Participants) | 94 | 93 | 99 | 97
  Absolute Change from Baseline at Month 6 | 18.1 (1.88) | 17.2 (1.87) | 15.4 (1.81) | 18.6 (1.85)
  Absolute Change from Baseline at Month 9: number analyzed (Participants) | 83 | 80 | 83 | 81
  Absolute Change from Baseline at Month 9 | 16.2 (193) | 14.7 (1.93) | 13.9 (1.88) | 16.3 (1.92)
  Absolute Change from Baseline at Month 12: number analyzed (Participants) | 95 | 92 | 98 | 96
  Absolute Change from Baseline at Month 12 | 18.9 (1.88) | 17.3 (1.88) | 16.4 (1.81) | 18.5 (1.85)

3. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) - Total Score
Description: The KOOS questionnaire assesses the participant's opinion about their osteoarthritis and associated problems. It consists of 5 subscales: pain, symptoms, activities of daily living (ADL) function, sport and recreation function, and knee related quality of life (QoL). The KOOS has 42 items across all subscales and response options are given on a 5-point Likert scale where 0 = no problems and 4 = extreme problems. The sum of subscale scores is transformed to a scale ranging from 0 to 100 with 0 indicating extreme symptoms and 100 indicating no symptoms. A negative value means that pain has worsened from what it was at baseline, while a positive value means that pain has improved from baseline.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: This analysis includes participants who successfully completed this assessment at the indicated post-baseline study visit. Some participants withdrew from the study prior to study completion and some attended study visits but did not complete each study assessment correctly. This analysis includes participants who had complete information for each subscale of the KOOS questionnaire, allowing for calculation of the total KOOS score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 100 | 95 | 109 | 101
score on a scale
  Change from Baseline at Month 1 | 14.48 (14.95) | 14.34 (12.40) | 11.14 (12.47) | 17.70 (14.65)
  Change from Baseline at Month 3: number analyzed (Participants) | 97 | 95 | 104 | 101
  Change from Baseline at Month 3 | 18.63 (15.32) | 16.30 (16.02) | 13.85 (14.36) | 17.21 (16.97)
  Change from Baseline at Month 6: number analyzed (Participants) | 91 | 88 | 96 | 97
  Change from Baseline at Month 6 | 18.39 (16.96) | 17.53 (16.23) | 15.62 (14.66) | 17.44 (17.47)
  Change from Baseline at Month 9: number analyzed (Participants) | 82 | 78 | 82 | 81
  Change from Baseline at Month 9 | 14.17 (18.87) | 13.36 (16.91) | 13.96 (15.83) | 116.30 (18.54)
  Change from Baseline at Month 12: number analyzed (Participants) | 95 | 89 | 96 | 94
  Change from Baseline at Month 12 | 18.52 (18.93) | 17.61 (19.70) | 17.49 (18.34) | 19.27 (18.54)

4. Secondary Outcome: Change in EuroQuality of Life (EQ-5D-3L) Index Score
Description: The EQ-5D-3L survey measures the severity of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participants will be asked to answer questions regarding these measures and to indicate their current experience on a scale from 1 to 3 (1 being "no problem" and 3 being "most extreme problem"). A sixth item asks participants to rate their current heath from 0 (worst imaginable) to 100 (best imaginable). The answers to these questions are converted into an index value based on the country respondents live in. Health state index scores typically range from less than 0 to 1, where 0 is a health state equivalent to death and 1 is perfect health. Positive values for the change from baseline score indicate improved health.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 100 | 101 | 111 | 100
score on a scale
  Absolute Change from Baseline at Month 1: number analyzed (Participants) | 100 | 100 | 111 | 100
  Absolute Change from Baseline at Month 1 | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01)
  Absolute Change from Baseline at Month 3: number analyzed (Participants) | 98 | 101 | 105 | 99
  Absolute Change from Baseline at Month 3 | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01)
  Absolute Change from Baseline at Month 6: number analyzed (Participants) | 94 | 93 | 98 | 96
  Absolute Change from Baseline at Month 6 | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01)
  Absolute Change from Baseline at Month 9: number analyzed (Participants) | 83 | 80 | 83 | 80
  Absolute Change from Baseline at Month 9 | 0.0 (0.02) | 0.1 (0.02) | 0.1 (0.02) | 0.1 (0.02)
  Absolute Change from Baseline at Month 12: number analyzed (Participants) | 95 | 92 | 97 | 95
  Absolute Change from Baseline at Month 12 | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01) | 0.1 (0.01)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Score
Description: The PROMIS-29 assesses seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. The PROMIS-29 scales are scored using a T-score metric method available at the Assessment Center website (http://assessmentcenter.net). A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Scores higher than 50 indicate more of the specific scale's construct, which may indicate a desirable or an undesirable outcome.
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
Population: This analysis includes participants who successfully completed this assessment at the indicated post-baseline study visit. Some participants withdrew from the study prior to study completion and some attended study visits but did not complete each study assessment correctly. Participants with incomplete responses are not included in the analysis for that domain.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 114 | 115 | 116 | 116
t-score
  Anxiety Score - Baseline | 47.1 (7.89) | 47.5 (7.79) | 47.1 (7.31) | 48.2 (8.69)
  Anxiety Score - Month 1: number analyzed (Participants) | 99 | 99 | 111 | 100
  Anxiety Score - Month 1 | 45.9 (7.46) | 45.4 (7.64) | 45.9 (7.73) | 45.4 (7.83)
  Anxiety Score - Month 3: number analyzed (Participants) | 98 | 100 | 104 | 100
  Anxiety Score - Month 3 | 45.1 (7.34) | 45.4 (7.91) | 45.4 (7.15) | 45.5 (7.67)
  Anxiety Score - Month 6: number analyzed (Participants) | 93 | 92 | 98 | 96
  Anxiety Score - Month 6 | 45.9 (7.45) | 45.8 (8.23) | 45.2 (7.51) | 45.3 (6.66)
  Anxiety Score - Month 9: number analyzed (Participants) | 81 | 80 | 83 | 81
  Anxiety Score - Month 9 | 46.1 (8.04) | 45.4 (7.94) | 44.9 (6.53) | 45.1 (6.88)
  Anxiety Score - Month 12: number analyzed (Participants) | 94 | 91 | 98 | 96
  Anxiety Score - Month 12 | 45.6 (8.10) | 45.3 (7.46) | 44.9 (7.25) | 45.2 (8.09)
  Depression Score - Baseline | 44.7 (5.70) | 45.0 (6.56) | 44.9 (6.34) | 45.6 (7.61)
  Depression Score - Month 1: number analyzed (Participants) | 99 | 99 | 111 | 101
  Depression Score - Month 1 | 44.3 (6.54) | 43.8 (6.19) | 44.9 (5.97) | 45.0 (6.92)
  Depression Score - Month 3: number analyzed (Participants) | 98 | 100 | 105 | 100
  Depression Score - Month 3 | 43.8 (5.56) | 44.0 (6.46) | 44.4 (5.88) | 446 (6.60)
  Depression Score - Month 6: number analyzed (Participants) | 93 | 92 | 98 | 96
  Depression Score - Month 6 | 43.9 (5.98) | 44.9 (6.50) | 44.0 (5.44) | 44.0 (5.38)
  Depression Score - Month 9: number analyzed (Participants) | 81 | 80 | 83 | 80
  Depression Score - Month 9 | 45.6 (6.99) | 45.2 (6.71) | 43.4 (5.03) | 44.1 (5.78)
  Depression Score - Month 12: number analyzed (Participants) | 94 | 91 | 98 | 96
  Depression Score - Month 12 | 44.5 (6.33) | 43.9 (6.01) | 44.3 (6.05) | 44.5 (6.65)
  Fatigue Score - Baseline: number analyzed (Participants) | 114 | 114 | 116 | 116
  Fatigue Score - Baseline | 46.8 (8.35) | 47.0 (8.29) | 47.7 (7.39) | 48.5 (8.92)
  Fatigue Score - Month 1: number analyzed (Participants) | 99 | 99 | 111 | 101
  Fatigue Score - Month 1 | 45.8 (8.94) | 45.8 (8.96) | 46.9 (8.45) | 46.2 (8.55)
  Fatigue Score - Month 3: number analyzed (Participants) | 98 | 99 | 105 | 100
  Fatigue Score - Month 3 | 45.0 (9.35) | 45.3 (8.50) | 46.0 (7.86) | 44.8 (8.50)
  Fatigue Score - Month 6: number analyzed (Participants) | 92 | 91 | 98 | 96
  Fatigue Score - Month 6 | 45.9 (9.52) | 46.1 (8.77) | 44.9 (8.57) | 45.1 (8.30)
  Fatigue Score - Month 9: number analyzed (Participants) | 81 | 80 | 83 | 80
  Fatigue Score - Month 9 | 46.7 (9.39) | 46.1 (8.98) | 47.1 (8.35) | 46.8 (9.70)
  Fatigue Score - Month 12: number analyzed (Participants) | 94 | 90 | 98 | 96
  Fatigue Score - Month 12 | 45.6 (9.09) | 45.2 (8.26) | 45.9 (8.66) | 45.3 (9.84)
  Pain Score - Baseline | 59.1 (6.06) | 58.6 (6.72) | 58.9 (5.58) | 60.4 (6.56)
  Pain Score - Month 1: number analyzed (Participants) | 97 | 99 | 111 | 100
  Pain Score - Month 1 | 53.6 (7.76) | 52.5 (6.82) | 54.8 (7.98) | 53.3 (7.81)
  Pain Score - Month 3: number analyzed (Participants) | 98 | 100 | 105 | 100
  Pain Score - Month 3 | 51.6 (8.17) | 52.1 (7.42) | 52.5 (7.86) | 53.5 (8.72)
  Pain Score - Month 6: number analyzed (Participants) | 92 | 92 | 98 | 97
  Pain Score - Month 6 | 51.5 (8.80) | 51.5 (8.00) | 51.9 (7.71) | 53.6 (7.67)
  Pain Score - Month 9: number analyzed (Participants) | 81 | 80 | 82 | 80
  Pain Score - Month 9 | 52.4 (8.55) | 52.3 (8.21) | 51.8 (8.14) | 53.2 (8.77)
  Pain Score - Month 12: number analyzed (Participants) | 94 | 91 | 98 | 96
  Pain Score - Month 12 | 51.5 (8.47) | 50.8 (8.23) | 51.2 (8.26) | 52.7 (8.48)
  Physical Function Score - Baseline: number analyzed (Participants) | 113 | 115 | 116 | 116
  Physical Function Score - Baseline | 39.3 (5.30) | 40.3 (5.80) | 38.8 (4.04) | 38.3 (5.10)
  Physical Function Score - Month 1: number analyzed (Participants) | 97 | 98 | 111 | 100
  Physical Function Score - Month 1 | 43.0 (7.30) | 43.6 (5.48) | 41.9 (6.07) | 43.3 (6.12)
  Physical Function Score - Month 3: number analyzed (Participants) | 97 | 98 | 105 | 101
  Physical Function Score - Month 3 | 44.9 (7.77) | 44.3 (5.84) | 43.8 (6.81) | 42.9 (7.03)
  Physical Function Score - Month 6: number analyzed (Participants) | 92 | 91 | 98 | 96
  Physical Function Score - Month 6 | 44.5 (7.33) | 45.2 (6.72) | 44.2 (6.59) | 43.0 (6.15)
  Physical Function Score - Month 9: number analyzed (Participants) | 80 | 80 | 83 | 81
  Physical Function Score - Month 9 | 43.0 (7.32) | 44.6 (6.60) | 44.4 (7.17) | 43.0 (6.76)
  Physical Function Score - Month 12: number analyzed (Participants) | 93 | 90 | 98 | 96
  Physical Function Score - Month 12 | 44.4 (7.81) | 45.2 (7.20) | 44.8 (7.25) | 43.6 (6.84)
  Sleep Disturbance Score - Baseline: number analyzed (Participants) | 113 | 114 | 116 | 116
  Sleep Disturbance Score - Baseline | 48.9 (7.00) | 49.7 (7.74) | 50.1 (7.92) | 50.2 (8.07)
  Sleep Disturbance Score - Month 1: number analyzed (Participants) | 99 | 99 | 111 | 101
  Sleep Disturbance Score - Month 1 | 47.2 (7.48) | 48.4 (7.63) | 48.3 (8.66) | 49.2 (7.91)
  Sleep Disturbance Score - Month 3: number analyzed (Participants) | 97 | 99 | 104 | 101
  Sleep Disturbance Score - Month 3 | 47.3 (7.94) | 48.3 (7.85) | 47.8 (7.90) | 47.9 (8.18)
  Sleep Disturbance Score - Month 6: number analyzed (Participants) | 91 | 92 | 98 | 97
  Sleep Disturbance Score - Month 6 | 48.6 (8.31) | 48.9 (6.88) | 48.1 (7.89) | 48.9 (7.38)
  Sleep Disturbance Score - Month 9: number analyzed (Participants) | 80 | 80 | 83 | 80
  Sleep Disturbance Score - Month 9 | 48.9 (7.50) | 48.5 (7.35) | 48.9 (7.77) | 47.9 (8.17)
  Sleep Disturbance Score - Month 12: number analyzed (Participants) | 93 | 90 | 98 | 96
  Sleep Disturbance Score - Month 12 | 47.8 (8.42) | 49.0 (7.02) | 48.7 (8.05) | 48.8 (8.08)
  Social Roles and Activities Score - Baseline | 49.5 (8.24) | 47.9 (8.33) | 48.2 (7.18) | 46.9 (7.53)
  Social Roles and Activities Score - Month 1: number analyzed (Participants) | 97 | 99 | 109 | 100
  Social Roles and Activities Score - Month 1 | 52.1 (8.69) | 51.6 (7.83) | 51.0 (7.65) | 51.5 (8.30)
  Social Roles and Activities Score - Month 3: number analyzed (Participants) | 98 | 100 | 105 | 101
  Social Roles and Activities Score - Month 3 | 54.4 (9.36) | 53.3 (8.18) | 52.4 (8.25) | 51.6 (9.00)
  Social Roles and Activities Score - Month 6: number analyzed (Participants) | 92 | 92 | 98 | 97
  Social Roles and Activities Score - Month 6 | 53.1 (8.77) | 52.7 (8.32) | 52.3 (8.15) | 52.0 (8.56)
  Social Roles and Activities Score - Month 9: number analyzed (Participants) | 81 | 80 | 82 | 80
  Social Roles and Activities Score - Month 9 | 53.6 (9.02) | 52.6 (8.41) | 52.8 (8.33) | 52.4 (8.47)
  Social Roles and Activities Score - Month 12: number analyzed (Participants) | 94 | 91 | 98 | 96
  Social Roles and Activities Score - Month 12 | 53.3 (9.02) | 53.5 (8.51) | 53.6 (8.05) | 52.2 (8.30)

6. Secondary Outcome: Overall MRI Grade of Osteoarthritis
Description: An MRI grade of osteoarthritis was calculated by rating features viewed by MRI (such as cartilage loss) in terms of severity and extent. Total scores range from 0 to 69 with higher values indicating more severe osteoarthritis.
Time Frame: Baseline, Month 6, Month 12
Population: This analysis includes participants who successfully completed the MRI assessment at the indicated study visit. Some participants withdrew from the study prior to reaching study visits where the MRI was conducted. Some participants who attended the MRI visit were not able to hold still during the entire MRI and an accurate measurement could not be obtained.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
Number analyzed (Participants) | 103 | 107 | 108 | 101
score on a scale
  Baseline | 40.5 (6.19) | 39.7 (7.82) | 38.2 (7.77) | 38.9 (7.70)
  Month 6: number analyzed (Participants) | 95 | 93 | 99 | 98
  Month 6 | 40.4 (6.27) | 39.3 (7.55) | 38.3 (7.86) | 39.3 (7.88)
  Month 12: number analyzed (Participants) | 93 | 85 | 96 | 95
  Month 12 | 40.8 (6.01) | 39.8 (7.76) | 37.6 (7.81) | 39.0 (7.84)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time participants began receiving the study intervention until the Month 12 follow-up visit.
Arm/Group | Bone Marrow Derived MSCs | Adipose-derived MSCs | Umbilical Cord Tissue (UCT) MSCs | Corticosteroid Injection
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/109 | 0/116 | 0/108
Serious Adverse Events (participants affected / at risk) | 8/107 | 2/109 | 4/116 | 5/108
Other Adverse Events (participants affected / at risk) | 53/107 | 64/109 | 45/116 | 48/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Derived MSCs (N=107) | Adipose-derived MSCs (N=109) | Umbilical Cord Tissue (UCT) MSCs (N=116) | Corticosteroid Injection (N=108)
Metastatic breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 | 0 | 0
Angina pectoris (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0 | 0
Atrial fibrillation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Traumatic pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Ischemic stroke (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Migraine (Nervous system disorders) | 1 (1) | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1)
Hypertension urgency (Vascular disorders) | 1 (1) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bone Marrow Derived MSCs (N=107) | Adipose-derived MSCs (N=109) | Umbilical Cord Tissue (UCT) MSCs (N=116) | Corticosteroid Injection (N=108)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 25 | 30 | 28
Joint stiffness (Musculoskeletal and connective tissue disorders) | 13 | 6 | 8 | 8
Joint swelling (Musculoskeletal and connective tissue disorders) | 19 | 16 | 28 | 8
Post procedural contusion (Injury, poisoning and procedural complications) | 11 | 41 | 0 | 21
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 12 | 0 | 7
Procedural pain (Injury, poisoning and procedural complications) | 28 | 37 | 0 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03818737/Prot_SAP_000.pdf